CLINICAL TRIAL: NCT06782074
Title: Idiopathic Generalized Epilepsy: Cognitive, Emotional, Behavioral Functioning, and Quality of Life
Brief Title: Idiopathic Generalized Epilepsy Cognitive and Emotional Profile
Status: Recruiting | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Buzzi Children's Hospital, Milan, Italy (Unknown); University of Catanzaro, Italy (Unknown); ASST Rhodense, Rho, Milan, Italy (Unknown)
Responsible Party: Sponsor
Other Study IDs: IGE
Record Dates: First submitted 2024-12-06; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Epilepsy; Quality of Life; Neuropathology; Emotional Problem; Executive Dysfunction
MeSH Terms: conditions — Epilepsy | interventions — Neuropsychological Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: emotional and neuropsychological assessment — The tests for evaluating emotional-behavioral functioning and quality of life will be self-administered by the patient/caregiver during regular follow-up visits. The cognitive assessment will be conducted by the clinician using standardized tests.

SUMMARY:
The primary goal of the study is to explore the neurocognitive, emotional-behavioral functioning, and quality of life of adolescents with IGE, identifying key factors that affect their overall well-being.

The study involves participants and their caregivers completing standardized questionnaires. Additionally, clinical and anamnesic information will be collected to investigate the role of these variables on the emotional and executive functioning of the enrolled subjects

DETAILED DESCRIPTION:
The 2022 ILAE classification includes several types of idiopathic generalized epilepsy (IGE), including childhood absence epilepsy (CAE), adolescent absence epilepsy (JAE), juvenile myoclonic epilepsy (JME), and generalized tonic-clonic seizure epilepsy (GTCA). While neurocognitive development is generally normal, these conditions are often associated with mood disorders, ADHD, and learning disabilities. Prognostically, patients with IGE tend to experience negative social outcomes such as poor academic performance, increased risk of unintended pregnancies, and psychiatric or emotional problems. These conditions may involve a range of seizure types, including absence, myoclonic, and tonic-clonic seizures, with EEG showing generalized spikes of 2.5-5.5 Hz.

These epilepsy syndromes are typically responsive to medication, but polytherapy is often required for optimal seizure control. The likelihood of remission and the age of remission can vary between syndromes, and patients may transition from one IGE syndrome to another. In recent years, the focus of epilepsy treatment has shifted beyond seizure control to include psychological factors, aiming to improve the patient's overall health-related quality of life (HRQOL). Studies have shown that children with epilepsy have lower HRQOL compared to healthy controls or children with other chronic conditions. Factors influencing HRQOL include psychiatric comorbidities, psychosocial challenges, cognitive and executive functioning, as well as epilepsy-specific variables such as seizure frequency, duration, and medication side effects.

The primary goal of the study is to explore the neurocognitive, emotional-behavioral functioning, and quality of life of adolescents with IGE, identifying key factors that affect their overall well-being.

ELIGIBILITY:
Inclusion criteria:

Age between 11 and 18 years Diagnosis of idiopathic generalized epilepsy

Exclusion criteria:

Age under 11 years or over 18 years Structural or cryptogenic epilepsy Intellectual disability or borderline cognitive level Refusal to participate in the study Failure to obtain informed consent

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: All patients attending the participating clinical units during the 2-year study period will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
cognition in patients with IGE throughout standardized tool WISC IV Wechsler Intelligence Scale for Children - Fourth Edition) or WAIS IV Wechsler Adult Intelligence Scale | 1 year
  The study includes the administration of standardized tool (WISC IV or WAIS IV) to describe the cognitive profile of these patients . Minimum score 40 max 160, average score 100, higher scores mean a better performance
quality of life in patients with IGE throughout standardized questionnaire | 1 year
  The study wants to describe quality of life in patients with IGE using standardized questionaire Pediatric Quality of Life Inventory (PedsQL)epilepsy module (min score 0, max 100; higher scores reflect a better quality of life).
behavioral profile in patients with IGE throughout standardized questionnaire | 1 year
  The study aims to define the behavioral profile of patients with IGE using standardized questionnaire: Child Behavior Checklist CBCL (min 0 max 200 higher score worse emotional profile) ,SAFA Strumenti di Autovalutazione per Fanciulli e Adolescenti (Self-Assessment Tools for Children and Adolescents (score min 0 max 100 Higher scores indicate greater emotional or behavioral difficulties.
executive profile of patients with IGE using standardized questionnaire BRIEF 2 | 1 year
  The study aims to define the executive profile of patients with IGE using standardized questionnaire Behavior Rating Inventory of Executive Function, Second Edition BRIEF 2 (score min 0 max 160 Higher scores indicate greater executive function difficulties.)

SECONDARY OUTCOMES:
correlation between presence of neurodevelopmental comorbilities and quality of life using an ad hoc questionnaire | 1 year
  The secondary objective of this study is to examine the correlation between the presence or absence of neurodevelopmental comorbidities and the quality of life (QoL). To assess the possible presence of these comorbidities, an ad hoc questionnaire will be used, which investigates the presence of potential comorbidities.

OTHER OUTCOMES:
correlation between seizure frequency and qol using an ad hoc questionnaire | 1 year
  The secondary objective of this study is to examine the correlation between the frequency of epileptic seizures and the quality of life (QoL). The annual frequency of seizures will be determined through an ad hoc questionnaire completed by the clinician.
correlation between the use of antiseizure medication and quality of life using a standardized questionnaire | 1 year
  The secondary objective of this study is to examine the correlation between the use of antiepileptic therapy and the quality of life (QoL). The use of antiepileptic therapy will also be assessed as part of the study through an ad hoc questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No